CLINICAL TRIAL: NCT02754024
Title: Humeral Head Implants: Radiological and Clinical Evaluation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Werner Anderl (Other)
Responsible Party: Sponsor-Investigator, Werner Anderl, Member, Austrian Research Group for Regenerative and Orthopedic Medicine
Organization: Austrian Research Group for Regenerative and Orthopedic Medicine (Other)
Other Study IDs: HHI
Record Dates: First submitted 2016-04-21; First posted 2016-04-28 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Idiopathic Osteoarthritis; Posttraumatic Osteoarthritis; Humeral Head Necrosis; Instability Arthritis
Keywords: Stemless shoulder prosthesis
MeSH Terms: interventions — Arthroplasty, Replacement, Shoulder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Total shoulder arthroplasty (TSA): Replacement of humeral head and glenoid
  Interventions: Procedure: Total shoulder arthroplasty (TSA); Device: Eclipse™ (Arthrex Inc., Naples, FL, USA)
- Hemi shoulder arthroplasty (HSA): Replacement of humeral head only
  Interventions: Procedure: Hemi shoulder arthroplasty (HSA); Device: Eclipse™ (Arthrex Inc., Naples, FL, USA)

INTERVENTIONS:
Procedure: Total shoulder arthroplasty (TSA) — stemless humeral head implant: Eclipse™ (Arthrex Inc., Naples, FL, USA)
  Groups: Total shoulder arthroplasty (TSA)
Procedure: Hemi shoulder arthroplasty (HSA) — stemless humeral head implant: Eclipse™ (Arthrex Inc., Naples, FL, USA)
  Groups: Hemi shoulder arthroplasty (HSA)
Device: Eclipse™ (Arthrex Inc., Naples, FL, USA) — stemless humeral head implant

SUMMARY:
In the past years several shoulder reconstruction systems with different types of prostheses and fixation methods have been developed to improve shoulder arthroplasty, trying to cover a wide range of pathologies and revision situations. The aim of the present study is to report radiological and clinical outcome with a stemless shoulder implant with hollow screw fixation.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 85 years at time of surgery
* Patients with primary or secondary osteoarthritis of the shoulder

Exclusion Criteria:

* Patients with cuff tear arthropathy and axillary nerve lesions

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring hemi- or total shoulder arthroplasty
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2005-09; Primary Completion 2016-03 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
the Constant score | 5 years
  The Constant score is a validated outcome score assessing pain and function of the shoulder
Radiological assessment to determine radiolucent areas and osteolysis around the humeral head | 5 years

SECONDARY OUTCOMES:
the Constant score | Change from baseline to 2 years postimplantation
Radiological assessment to determine radiolucent areas and osteolysis around the humeral head | 2 years
the Constant score | Change from baseline to 5 years postimplantation
the Constant score | 10 years
Radiological assessment to determine radiolucent areas and osteolysis around the humeral head | 10 years
the Constant score | 15-20 years
Radiological assessment to determine radiolucent areas and osteolysis around the humeral head | 15-20 years

REFERENCES:
- [Derived] Heuberer PR, Brandl G, Pauzenberger L, Laky B, Kriegleder B, Anderl W. Radiological changes do not influence clinical mid-term outcome in stemless humeral head replacements with hollow screw fixation: a prospective radiological and clinical evaluation. BMC Musculoskelet Disord. 2018 Jan 22;19(1):28. doi: 10.1186/s12891-018-1945-6. PMID 29357861